CLINICAL TRIAL: NCT01146366
Title: Utility of Routine Cervical Mediastinoscopy in Clinically Staged T2N0M0 and Select T1N0M0 Non-Small Cell Lung Cancers by FDG-PET and CT Scans
Brief Title: Utility of Routine Cervical Mediastinoscopy in Clinical Stage I Non-Small Cell Lung Cancer (NSCLC)
Status: Completed | Type: Observational
Sponsor: Jennifer Bell (Other)
Collaborators: University of Virginia (Other); University of North Carolina (Other); Emory University (Other)
Responsible Party: Sponsor-Investigator, Jennifer Bell, Manager of Research, Cardiothoracic Surgery, Washington University School of Medicine
Organization: Washington University School of Medicine (Other)
Other Study IDs: 08-0020
Record Dates: First submitted 2010-06-10; First posted 2010-06-17 (Estimated); Last update posted 2014-12-11 (Estimated); Status verified 2014-12

CONDITIONS: Non-small Cell Lung Cancer
Keywords: Early stage lung cancer; Cervical mediastinoscopy; Observational study; clinical stage T2N0M0 and select T1N0M0 (suvMAX on FDG-PET of >/=10)
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
To prospectively look at the utility of routine cervical mediastinoscopy (lymph node biopsy) in patients with clinically staged T2N0M0 NSCLC, as well as patients with clinically staged T1N0M0 NSCLC with a high maxSUV of the primary tumor on PET imaging.

Hypothesis #1: The prevalence of mediastinal lymph node metastases detectable by cervical mediastinoscopy is sufficiently low (<10%) to not support the routine use of this test in the study population.

Hypothesis #2: The preoperative detection of occult(hidden) N2 lymph node metastases by cervical mediastinoscopy in patients with clinically staged T2N0M0 NSCLC or T1N0M0 NSCLC with maxSUV >10 on PET does not provide a survival benefit when compared to detection of occult N2 lymph node metastases at the time of thoracotomy using nodal dissection or systematic sampling.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must have proven or suspected clinical stage I NSCLC. Clinical stage IA (T1N0M0) patients are only allowed participation if the maxSUV of the primary tumor is >/=10. Clinical stage IB (T2N0M0) must be by size criterion only (i.e. the tumor must be > 3cm in size. Patients that have T2 tumors by visceral pleural involvement only are not eligible for the study).
2. Patients must be surgical candidates for at least a lobectomy or other anatomical resection (via either video-assisted thoracoscopic surgery, or open approach).
3. Patient must have an ECOG/Zubrod score of 0, 1 or 2.
4. Patients must not have undergone previous invasive mediastinal staging for this cancer.
5. Patients must not have a tracheostomy.
6. Patient must have a CT of the chest and upper abdomen or an FDG-PET scan performed within 60 days of enrollment to the study that confirms their clinical stage I status. Both scans must be performed, only one needs to be within 60 days of enrollment to the study.

Exclusion Criteria:

There are no separately noted exclusion criteria. All criteria are listed under inclusion.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients being evaluated by a thoracic surgeon for surgical resection of clinical stage I non-small cell lung cancer
Sampling Method: Non-Probability Sample
Enrollment: 111 (Actual)
Dates: Start 2008-01; Primary Completion 2014-10 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Prevalence of occult N2/3 metastases in the study population | After cervical mediastinoscopy is performed in all subjects, estimated completion of enrollment of all subjects is 12/2012.
  Prevalence of occult N2/3 metastases in the study population. This is the fraction of enrolled patients with N2/3 metastases detected by either mediastinoscopy or by systematic sampling/dissection.

SECONDARY OUTCOMES:
Sensitivity of cervical mediastinoscopy for clinically occult N2 metastases | After cervical mediastinoscopy is performed in all subjects, estimated completion of enrollment of all subjects is 12/2012.
  Sensitivity of cervical mediastinoscopy for clinically occult N2 metastases. This is the number of patients with positive mediastinoscopy divided by the total number with N2/3 disease detected by either mediastinoscopy or by systematic sampling/dissection.

CONTACTS AND LOCATIONS:
Overall Officials: Bryan F Meyers, MD, MPH, Principal Investigator — Washington University School of Medicine
Locations (4):
- United States (4):
  - Emory University, Atlanta, Georgia
  - Washington University School of Medicine, St Louis, Missouri
  - University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - University of Virginia Health System, Charlottesville, Virginia

REFERENCES:
- [Background] Meyers BF, Haddad F, Siegel BA, Zoole JB, Battafarano RJ, Veeramachaneni N, Cooper JD, Patterson GA. Cost-effectiveness of routine mediastinoscopy in computed tomography- and positron emission tomography-screened patients with stage I lung cancer. J Thorac Cardiovasc Surg. 2006 Apr;131(4):822-9; discussion 822-9. doi: 10.1016/j.jtcvs.2005.10.045. Epub 2006 Mar 2. PMID 16580440
- [Background] Reed CE, Harpole DH, Posther KE, Woolson SL, Downey RJ, Meyers BF, Heelan RT, MacApinlac HA, Jung SH, Silvestri GA, Siegel BA, Rusch VW; American College of Surgeons Oncology Group Z0050 trial. Results of the American College of Surgeons Oncology Group Z0050 trial: the utility of positron emission tomography in staging potentially operable non-small cell lung cancer. J Thorac Cardiovasc Surg. 2003 Dec;126(6):1943-51. doi: 10.1016/j.jtcvs.2003.07.030. PMID 14688710
- [Background] Hammoud ZT, Anderson RC, Meyers BF, Guthrie TJ, Roper CL, Cooper JD, Patterson GA. The current role of mediastinoscopy in the evaluation of thoracic disease. J Thorac Cardiovasc Surg. 1999 Nov;118(5):894-9. doi: 10.1016/s0022-5223(99)70059-0. PMID 10534695
- [Background] Gonzalez-Stawinski GV, Lemaire A, Merchant F, O'Halloran E, Coleman RE, Harpole DH, D'Amico TA. A comparative analysis of positron emission tomography and mediastinoscopy in staging non-small cell lung cancer. J Thorac Cardiovasc Surg. 2003 Dec;126(6):1900-5. doi: 10.1016/s0022-5223(03)01036-5. PMID 14688703
- [Background] Cerfolio RJ, Bryant AS, Ohja B, Bartolucci AA. The maximum standardized uptake values on positron emission tomography of a non-small cell lung cancer predict stage, recurrence, and survival. J Thorac Cardiovasc Surg. 2005 Jul;130(1):151-9. doi: 10.1016/j.jtcvs.2004.11.007. PMID 15999056
- [Derived] Fernandez FG, Kozower BD, Crabtree TD, Force SD, Lau C, Pickens A, Krupnick AS, Veeramachaneni N, Patterson GA, Jones DR, Meyers BF. Utility of mediastinoscopy in clinical stage I lung cancers at risk for occult mediastinal nodal metastases. J Thorac Cardiovasc Surg. 2015 Jan;149(1):35-41, 42.e1. doi: 10.1016/j.jtcvs.2014.08.075. Epub 2014 Sep 17. PMID 25439769